CLINICAL TRIAL: NCT03236779
Title: A Comparative Study of Two Dry Needling Interventions for Plantar Heel Pain: A Randomized Clinical Trial
Brief Title: A Comparative Study of Two Dry Needling Interventions for Plantar Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Universidad San Jorge (Other); Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, ZAID AL BOLOUSHI, PhD student, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALBOLOUSHI
Record Dates: First submitted 2017-07-25; First posted 2017-08-02 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Plantar Fascitis; Myofacial Pain Syndromes; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Facial Neuralgia; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: This study is a prospective, two parallel-groups (participant) randomized controlled trial with blinded outcome assessment at baseline, and at 4, 8, 12, 26 and 52 weeks. The study flow chart shown in Figure 1 conforms to the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines for nonpharmacological studies
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants who fulfill the inclusion criteria will receive the standardized oral and written information, and, once they consent to participate in the trial, will be randomized in a block system by blocks of 10 patients. Allocation to the groups will be achieved using a computer program (Randomizer, https://www.randomizer.org/) generated a random patient file numbers sequence by a third person not involved in the study from the file section in Kuwait. This person will be responsible for guarding the envelope with the information of the randomization. The envelopes will be closed until the moment of the intervention to maintain the blinding. This professional also will ask the patients for informed consent. The consent form is recruited upon the ethical medical committee at the ministry of health in the state of Kuwait.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (DN) arm (Experimental): Once the clinician locates the MTrP, he will insert the needle over it and he will do a quick entry of the needle. The chosen technique to manipulate the needle will be Hong technique, which consist of quick entry and exit of the needle (fast in/fast out) to get local twitch response (LTR), it will be repeated 5 times with a rhythmic movement of 1Hz/sec. LTRs will be counted and registered.
  Interventions: Other: dry needling
- Percutaneous needle electrolysis (PNE) arm (Active Comparator): The electrotherapy equipment used (Enraf) produces a continuous galvanic current through the cathode (modified electrosurgical scalpel with the needle) while the patient holds the anode (handheld electrode). Once the needle have reach the relevant treatment area, a continuous current of 3 pulses at an intensity of 3, 1.5 mA for 5 seconds conveyed to the muscle will be applied. It will be done exactly the same way as in the DN group with the only difference that the needle will be transmitting the electrical current.
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — The electrotherapy equipment used (Enruf) produces a continuous galvanic current through the cathode (modified electrosurgical scalpel with the needle) while the patient holds the anode (handheld electrode) (42). Once the needle have reach the relevant treatment area, a continuous current of 3 pulses at an intensity of 3 1.5 mA for 5 seconds conveyed to the muscle will be applied.
  Other Names: Percutaneous needle electrolysis

SUMMARY:
This is a clinical trial that will be done in the state of Kuwait, at the physical rehabilitation medicine hospital. the participants will be recruited from all over Kuwait, there is a clinical registry upon the ethical committee in Kuwait assigned by the ministry of health.

DETAILED DESCRIPTION:
Physical therapy approaches continue evolving. During the last years, minimally invasive techniques such as percutaneous needle electrolysis (PNE) was being developed, obtaining promising results for tendon pathology. PNE technique is a minimally invasive treatment that consists of an application of a galvanic electrolytic current that causes a controlled local inflammatory process in the target tissue. This allows for phagocytosis and the subsequent regeneration of the affected tissue. Nowadays, PNE is being used in clinical practice to manage MTrP, but there are no studies supporting that they have an additional beneficial effect over DN.

From a biological point of view, it seems reasonable to ascertain that a patient will obtain benefits thanks to the mechanical effects provided by the needle and that patients may benefit more if the electrolysis effect is added to the mechanical stimuli provided by the needle. Therefore, the aim of this randomized controlled study is to compare the effectiveness of DN versus PNE for the level of pain in patients suffering from PHP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PHP in accordance with the Clinical Guidelines linked to the International Classification of Function, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association
* Age greater than 21 years according to the Kuwaiti law.
* History of plantar heel pain for greater than one month.
* Walking 50 meters without any support
* Having MTPs on initial physical examination on plantar and calf muscles
* Accepting to be treated by a male physiotherapist.
* Capacity to understand the study and the informed consent, as well as having signed the document.

Exclusion Criteria:

* - Needle phobia
* Allergy from needles or hypersensitivity to metals
* Presence of coagulopathy or use of anticoagulants
* Presence of peripheral arterial vascular disease
* Pregnancy
* Dermatological disease with the dry needling area
* The presence of a chronic medical condition that might preclude participation in the study such as malignancy, systemic inflammatory disorders (e.g. psoriatic arthritis, ankylosing spondylitis, septic arthritis), neurological diseases, polyneuropathy, mononeuropathy.
* Treatment of plantar heel pain with needling or acupuncture during last 4 weeks.
* A history of injection therapy in the heel in the previous three months.
* Previous history of foot surgery or fracture.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Medicine and rehabilitation Kuwait, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No
ACCORDING TO THE LAW AND REGULATIONS FROM THE ETHICAL COMMITTEE IN KUWAIT. I CAN'T SHARE THE NAME OF THE PATIENTS, THEIR CONTACT OR ID. OTHER DATA WHICH ARE RELATED TO THE STUDY I CAN SHARE.

REFERENCES:
- [Derived] Fernandez D, Al-Boloushi Z, Bellosta-Lopez P, Herrero P, Gomez M, Calvo S. Cost-Effectiveness of Two Dry Needling Interventions for Plantar Heel Pain: A Secondary Analysis of an RCT. Int J Environ Res Public Health. 2021 Feb 12;18(4):1777. doi: 10.3390/ijerph18041777. PMID 33673068
- [Derived] Al-Boloushi Z, Gomez-Trullen EM, Arian M, Fernandez D, Herrero P, Bellosta-Lopez P. Comparing two dry needling interventions for plantar heel pain: a randomised controlled trial. BMJ Open. 2020 Aug 20;10(8):e038033. doi: 10.1136/bmjopen-2020-038033. PMID 32819949
- [Derived] Al-Boloushi Z, Gomez-Trullen EM, Bellosta-Lopez P, Lopez-Royo MP, Fernandez D, Herrero P. Comparing two dry needling interventions for plantar heel pain: a protocol for a randomized controlled trial. J Orthop Surg Res. 2019 Jan 25;14(1):31. doi: 10.1186/s13018-019-1066-4. PMID 30683124

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dry Needling (DN) Arm | Percutaneous Needle Electrolysis (PNE) Arm
Started | 51 | 51
Completed | 38 | 30
Not Completed | 13 | 21
Not completed — Lost to Follow-up | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dry Needling (DN) Arm | Percutaneous Needle Electrolysis (PNE) Arm | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.9) | 48.1 (8.8) | 48.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 51 | 51 | 102
Region of Enrollment [Count of Participants; unit: Participants]
  Kuwait | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Foot Health Status Questioner (FHSQ) PAIN
Description: Participants will complete the FHSQ at baseline and at 4, 8, 12, 26, and 52 weeks post-treatment. The FHSQ consists of 13 questions reflecting fourfoot health-related domains: pain (4 questions), function (4 questions), footwear (3 questions), and general foot health (2 questions). Individual item scores will then be re-coded, tabulated, and finally transformed to a scale ranging from 0 to 100 for each of the four domains. Greater scores reflect better foot health and quality of life. The FHSQ has been validated and has been used in similar trials that have evaluated the effectiveness of different interventions for plantar heel pain
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dry Needling (DN) Arm | Percutaneous Needle Electrolysis (PNE) Arm
Number analyzed (Participants) | 51 | 51
score on a scale
  baseline | 38.8 (18.8) | 40.4 (21.9)
  4 weeks | 73.4 (27.7) | 71.9 (25.7)
  8 weeks | 70.1 (28.4) | 67.4 (26.8)
  12 weeks | 66.8 (24.8) | 63.6 (26.8)
  26 weeks | 68.8 (25.3) | 67.1 (27.1)
  52 weeks | 68.4 (25.1) | 73.1 (29.0)

2. Secondary Outcome: VAS Maximum
Description: Participants will complete the visual analogue scale (VAS) before each treatment session, considering the level of pain they have just before start the treatment session and the highest level of pain they have had during the last 48 hours. The exact words of the questions will be: 1) what is the level of pain, as average, you have feel during last 48 hours?; and 2) what is the maximum level of pain you have feel during last 48 hours? Participants will be explained that a score of 0 indicates the absence of pain whereas a score of 10 represents the maximum tolerable pain. The VAS is widely used and is valid and reliable
Time Frame: 1st session (baseline), 2nd session (week 2), 3rd session (week 3), 4th session (week 4)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VAS DN; VAS PNE: the average and maximum level of pain over the past 48 hours using the visual analogue scale (VAS). Participants were explained that a score of 0 indicated the absence of pain whereas a score of 10 represented the maximum tolerable pain
Arm/Group | VAS DN | VAS PNE
Number analyzed (Participants) | 51 | 51
units on a scale
  baseline 1st session | 7.6 (2.0) | 7.5 (2.3)
  2nd session | 6.2 (2.3) | 5.5 (2.9)
  3rd session | 5.4 (2.6) | 5.3 (3.1)
  4th session | 4.9 (2.9) | 4.5 (3.0)

3. Secondary Outcome: The Quality of Life (QoL) Will be Assessed With the EuroQoL-5 Dimensions (EQ-5D)
Description: The EQ-5D-5L self-report questionnaire is a descriptive system with five questions, each representing one dimension of health-related QoL, that is, mobility, self-care, daily activities, pain/discomfort and depression/anxiety. Each dimension can be rated on five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Scoring is based on a 0 to 100% scale, where 100% represent the best QoL.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, 26 weeks, 52 weeks"
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dry Needling (DN) Arm | Percutaneous Needle Electrolysis (PNE) Arm
Number analyzed (Participants) | 51 | 51
units on a scale
  baseline | 0.63 (0.23) | 0.67 (0.22)
  4 weeks | 0.78 (0.22) | 0.76 (0.24)
  8 weeks | 0.72 (0.23) | 0.74 (0.23)
  12 weeks | 0.64 (0.30) | 0.70 (0.27)
  26 weeks | 0.65 (0.29) | 0.73 (0.27)
  52 weeks | 0.66 (0.27) | 0.77 (0.25)

4. Primary Outcome: Foot Health Status Questioner (FHSQ) PAIN
Description: as for outcome 1
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dry Needling (DN) Arm | Percutaneous Needle Electrolysis (PNE) Arm
Number analyzed (Participants) | 51 | 51
score on a scale
  baseline | 38.8 (18.8) | 40.4 (21.9)
  4 weeks | 73.4 (27.7) | 71.9 (25.7)
  8 weeks | 70.1 (28.4) | 67.4 (26.8)
  12 weeks | 66.8 (24.8) | 63.6 (26.8)
  26 weeks | 68.8 (25.3) | 67.1 (27.1)
  52 weeks | 68.4 (25.1) | 73.1 (29.0)

ADVERSE EVENTS:
Time Frame: 1 year follow up
Description: Unable to tolerate pain of the treatment
Groups:
- Dry Needling: Once the clinician located the MTrP, the needle was inserted over the same and a rapid needle entry was performed. The chosen technique for manipulating the needle was the technique described by Hong, which consists of a rapid needle entry and exit (fast in/fast out), in order to obtain a local twitch response, lasting 5 seconds employing a rhythmic movement at approximately 1Hz/sec (5 entries).
- Percutaneous Needle Electrolysis: The electrotherapy equipment used (Physio Invasiva, PRIM Fisioterapia, Spain) produced a continuous galvanic current through the cathode while the patient held a hand-held anode.18 Once the needle reached the relevant treatment area, this was needled in exactly the same manner as in the dry needling group, with the only difference being that the needle was transmitting an electrical current with an intensity of 1.5 mA (intensity was adapted to patient´s characteristics according to their pain tolerance).
Arm/Group | Dry Needling | Percutaneous Needle Electrolysis
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 9/51 | 14/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dry Needling (N=51) | Percutaneous Needle Electrolysis (N=51)
unable to tolerate pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (14) — Unable to tolerate pain of the treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03236779/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03236779/Prot_SAP_001.pdf